CLINICAL TRIAL: NCT00822094
Title: Phase IIB, Multicenter, Randomized, Open-Label Trial Of CPX-351 (Cytarabine : Daunorubicin) Liposome Injection Versus Intensive Salvage Therapy In Adult Patients ≤ 65 Years Old With AML In First Relapse Following An Initial CR > 1 Month Duration
Brief Title: Trial of CPX-351 in Adult Patients With First Relapse Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLTR0308-205
Record Dates: First submitted 2009-01-12; First posted 2009-01-14 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute; Myeloid; Leukemia; Adult; First; Relapse; AML; Acute Myelogenous leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute; Acute myelocytic leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Recurrence; Leukemia, Myeloid | interventions — CPX-351

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPX-351 (Arm A) (Experimental): First induction: 100 units/m2 on Days 1, 3, and 5 by 90-minute IV infusion Second induction: 100 units/m2 on Days 1 and 3 by 90-minute IV infusion Consolidation(s): 100 units/m2 on Days 1 and 3 by 90-minute IV infusion
  Interventions: Drug: CPX-351
- Salvage Therapy (Arm B) (Active Comparator): First induction: Investigator's choice salvage therapy administered according to local practice Second induction: Investigator's choice salvage therapy administered according to local practice Consolidation(s): Investigator's choice consolidation therapy administered according to local practice
  Interventions: Drug: Intensive Salvage Therapy

INTERVENTIONS:
Drug: CPX-351
  Arms: CPX-351 (Arm A)
Drug: Intensive Salvage Therapy
  Arms: Salvage Therapy (Arm B)

SUMMARY:
The study investigates if CPX-351 will be a) more effective than the standard intensive salvage AML treatment and b) more tolerable than the standard intensive salvage treatment regimens.

The study compares the investigational product CPX-351 vs the standard intensive salvage treatment for first relapse AML patients.

DETAILED DESCRIPTION:
This study is a randomized, open-label, parallel-arm, fixed-dose, standard therapy controlled Phase IIB trial. Study enrollment duration is expected to be approximately 12-18 months. On entry, patients are randomized to receive either CPX-351 or intensive first salvage treatment.

Patients are stratified to balance the likelihood of obtaining a CR and the duration of CR between the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and voluntarily sign an informed consent form
* Age ≥18 and ≤65 years at the time of relapse
* Pathological confirmation of relapsed AML after initial CR of >1 month duration
* Eastern Cooperative Oncology Group (ECOG) performance status 0- 2
* Able to adhere to the study visit schedule and other protocol requirements
* Laboratory values fulfilling the following:

  * Serum creatinine < 2.0 mg/dL
  * Serum total bilirubin < 2.0 mg/dL
  * Serum alanine aminotransferase or aspartate aminotransferase <3xULN Note: If elevated liver enzymes are related to disease; contact medical monitor to discuss.
* Cardiac ejection fraction > 50% by echocardiography or MUGA scan
* All men and women must agree to practice effective contraception during the study period and for 3 months afterward if not otherwise documented to be infertile.

Exclusion Criteria:

* Patients with active second malignancies are excluded. Patients with second malignancies in remission may be eligible if there is no clinical evidence of active disease, documented by imaging, with tumor marker studies, etc., at screening. Patients maintained on long-term non-chemotherapy treatment, e.g., hormonal therapy, are eligible. In all cases, the second malignancy and its non-chemotherapy treatment must not interfere with the investigators ability to assess the safety or efficacy of the study treatment
* Patients with acute promyelocytic leukemia [t(15;17)]
* Total lifetime anthracycline exposure exceeding the equivalent of 368 mg/m2 of daunorubicin (or equivalent) prior to start of study therapy
* Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent obtaining informed consent
* Administration of any antineoplastic therapy within 4 weeks of therapy; intended to treat first relapse. In the event of rapidly proliferative disease use of hydroxyurea is permitted until 24 hours before the start of study treatment
* Clinical evidence of active CNS leukemia
* Patients with history of and/or current evidence of myocardial impairment (e.g. cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, and congestive heart failure) resulting in New York Heart Association Class III or IV staging
* Active and uncontrolled infection. Patients with a bacterial infection receiving treatment with antibiotics may be entered into the study if they are afebrile and hemodynamically stable for >72 hrs.
* Current evidence of invasive fungal infection (blood or tissue culture); active hepatitis C infection or known HIV infection
* Hypersensitivity to cytarabine, daunorubicin or liposomal products
* History of Wilson's disease or other copper-related disorder
* Patients with a history of severe toxicity related to receiving conventional dose cytarabine in first line treatment (approximately 100mg/m2/d for <7 days) are excluded. Patients who experienced unacceptable toxicities while receiving high dose cytarabine (approximately 3000mg/m2 for 6 doses) will not be treated again with the same regimen, but could be randomized to treatment with conventional dose cytarabine regimens where the risk of major toxicity is less.
* Woman who are pregnant or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kolitz, MD, Principal Investigator — North Shore University Hospital
Locations (42):
- United States (31):
  - Arizona Cancer Center, Tucson, Arizona
  - UCLA, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UC Davis Cancer Center, Sacramento, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Northwestern University Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center Section of Hematology/Oncology, Chicago, Illinois
  - St. Francis Cancer Center, Beech Grove, Indiana
  - University of Louisville Brown Cancer Center, Louisville, Kentucky
  - Maine General Medical Center Harold Alfond Center for Cancer Care, Waterville, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - St. Louis University Medical Center, St Louis, Missouri
  - The Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - North Shore LIJ Center for Advanced Medicine Monter Cancer Center, Lake Success, New York
  - Weil Cornell Medical Center, New York, New York
  - New York Medical College, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Blumenthal Cancer Center/Mecklenburg Medical Group, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Jewish Hospital of Cincinatti, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Oncology and Hematology at Lehigh Valley, Bethlehem, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - UTMB Comprehensive Cancer Center, Galveston, Texas
  - M.D. Anderson Cancer Center, Houston, Texas
  - Joe Arrington Cancer Center, Lubbock, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Cancer Therapy and Research Center at The University of TX Health Science Center, San Antonio, Texas
  - Intermountain LDS Hospital, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Vancouver General Hospital/ British Columbia Cancer Agency, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
- France (4):
  - Service des Maladies du Sang CHU de Lille, Hopital Claude Huriez, Lille
  - Service des Maladies du Sang Hopital Haut-Leveque, Pessac
  - Service d'Hématologie CHU Toulouse-Hôpital Purpan, Toulouse
  - Service d'Hématologie et Médecine Interne CHU de Nancy-Hôpital de Brabois, Vandœuvre-lès-Nancy
- Poland (5):
  - Klinika Hematologii i Transplantologii, Gdansk
  - Wojewódzki Szpital Specjalistyczny im. M. Kopernika, Lodz
  - Oddział Hematologii, Opole
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Akademia Medyczna we Wroclawlu, Wroclaw

RESULTS

PARTICIPANT FLOW:
Groups:
- CPX-351: First induction: 100 units/m2 on Days 1, 3, and 5 by 90-minute IV infusion Second induction: 100 units/m2 on Days 1 and 3 by 90-minute IV infusion Consolidation(s): 100 units/m2 on Days 1 and 3 by 90-minute IV infusion
- Salvage Therapy: First induction: Investigator's choice salvage therapy administered according to local practice Second induction: Investigator's choice salvage therapy administered according to local practice Consolidation(s): Investigator's choice consolidation therapy administered according to local practice
Period: Overall Study
Arm/Group | CPX-351 | Salvage Therapy
Started | 81 | 45
Completed | 37 | 20
Not Completed | 44 | 25

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
  One subject in the Salvage Therapy arm was randomized and withdrew consent prior to treatment, and therefore was excluded from the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | CPX-351 | Salvage Therapy | Total
Number analyzed (Participants) | 81 | 44 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (11.57) | 51.8 (11.54) | 50.2 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 25 | 68
  Male | 38 | 19 | 57

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Surviving at 1 Year
Description: The proportion of subjects surviving at 1 year was evaluated separately for each arm by the number of subjects alive at 1 year divided by the total number of subjects.
Time Frame: Up to 1 year from randomization
Population: Efficacy Evaluable Analysis Set - All randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-351 | Salvage Therapy
Number analyzed (Participants) | 81 | 44
Participants | 29 | 12

2. Secondary Outcome: Complete Remission Rate
Time Frame: Following 1st induction, following 2nd induction if applicable
Population: Efficacy Evaluable Analysis Set: All randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-351 | Salvage Therapy
Number analyzed (Participants) | 81 | 44
Participants | 30 | 14

3. Secondary Outcome: Event Free Survival
Description: Progression EFS median
Time Frame: Up to 1 year from randomization
Population: Efficacy Evaluable Analysis Set: All randomized participants who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CPX-351 | Salvage Therapy
Number analyzed (Participants) | 81 | 44
days | 75 [43 to 128] | 43 [24 to 70]

4. Secondary Outcome: Remission Duration
Description: Remission duration was measured from the time the criteria for CR were first met until the first date that disease relapse was objectively documented or until subject death.
Time Frame: Following achievement of CR and up to 1 year from randomization
Population: Efficacy Evaluable Analysis Set: All randomized participants who received at least one dose of study medication.
Measure: Median (Full Range); unit: days
Arm/Group | CPX-351 | Salvage Therapy
Number analyzed (Participants) | 81 | 44
days | 301 [35 to 345] | 259 [47 to 354]

5. Secondary Outcome: Rate of Aplasia
Description: Patients with Aplasia During Study
Time Frame: Up to 1 year from randomization
Population: Efficacy Evaluable Analysis Set: All randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-351 | Salvage Therapy
Number analyzed (Participants) | 81 | 44
Participants | 62 | 24

6. Secondary Outcome: Rate of Stem Cell Transplant
Description: Number of patients transferred for stem cell transplant
Time Frame: Up to 1 year from randomization
Population: Efficacy Evaluable Analysis Set: All randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-351 | Salvage Therapy
Number analyzed (Participants) | 81 | 44
Participants | 38 | 21

ADVERSE EVENTS:
Time Frame: Continually assessed during Treatment Period and recorded and reported any new serious adverse events (up to 30 days after completion of Treatment Period)
Description: Safety Population: All randomized participants who received at least one dose of study medication.
Arm/Group | CPX-351 | Salvage Therapy
Serious Adverse Events (participants affected / at risk) | 53/81 | 22/44
Other Adverse Events (participants affected / at risk) | 81/81 | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CPX-351 (N=81) | Salvage Therapy (N=44)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Bone Marrow Necrosis (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 7 | 2
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 1
Conjunctival Haemorrhage (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Neutropenic Colitis (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Chest Pain (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Disease Progression (General disorders) | 0 | 1
Extravasation (General disorders) | 1 | 0
Mucosal Inflammation (General disorders) | 1 | 0
Multi-Organ Failure (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Sudden Cardiac Death (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 11 | 6
Catheter Site Infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Fungaemia (Infections and infestations) | 0 | 1
Gastrointestinal Bacterial Infection (Infections and infestations) | 1 | 0
Herpes Zoster Disseminated (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 2
Pneumonia Fungal (Infections and infestations) | 0 | 1
Pseudomonas Infection (Infections and infestations) | 0 | 1
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 8 | 1
Septic Shock (Infections and infestations) | 4 | 0
Sinusitis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Ejection Fraction Decreased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 2 | 0
Subclavian Vein Thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CPX-351 (N=81) | Salvage Therapy (N=44)
Anaemia (Blood and lymphatic system disorders) | 5 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 41 | 13
Lymphadenopathy (Blood and lymphatic system disorders) | 7 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3
Pericardial Effusion (Cardiac disorders) | 5 | 1
Tachycardia (Cardiac disorders) | 15 | 7
Abdominal Discomfort (Gastrointestinal disorders) | 5 | 2
Abdominal Distension (Gastrointestinal disorders) | 13 | 2
Abdominal Pain (Gastrointestinal disorders) | 17 | 9
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 34 | 12
Diarrhoea (Gastrointestinal disorders) | 31 | 26
Dry Mouth (Gastrointestinal disorders) | 5 | 3
Dyspepsia (Gastrointestinal disorders) | 8 | 5
Flatulence (Gastrointestinal disorders) | 6 | 0
Haemorrhoids (Gastrointestinal disorders) | 4 | 3
Mouth Haemorrhage (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 44 | 23
Oral Pain (Gastrointestinal disorders) | 4 | 3
Stomatitis (Gastrointestinal disorders) | 8 | 6
Vomiting (Gastrointestinal disorders) | 35 | 16
Asthenia (General disorders) | 11 | 9
Catheter Site Erythema (General disorders) | 7 | 4
Catheter Site Pain (General disorders) | 14 | 3
Chest Pain (General disorders) | 6 | 1
Chills (General disorders) | 24 | 10
Fatigue (General disorders) | 33 | 16
Mucosal Inflammation (General disorders) | 15 | 9
Oedema Peripheral (General disorders) | 34 | 11
Pain (General disorders) | 9 | 4
Pyrexia (General disorders) | 24 | 13
Drug Hypersensitivity (Immune system disorders) | 4 | 4
Bacteraemia (Infections and infestations) | 4 | 3
Cellulitis (Infections and infestations) | 8 | 4
Pneumonia (Infections and infestations) | 11 | 4
Urinary tract infection bacterial (Infections and infestations) | 0 | 3
Allergic Transfusion Reaction (Injury, poisoning and procedural complications) | 5 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 4 | 3
Transfusion Reaction (Injury, poisoning and procedural complications) | 3 | 6
Weight Decreased (Investigations) | 5 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 26 | 15
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 3
Hypnoatraemia (Metabolism and nutrition disorders) | 4 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 7 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 2
Dizziness (Nervous system disorders) | 16 | 5
Dysgeusia (Nervous system disorders) | 4 | 5
Headache (Nervous system disorders) | 23 | 15
Peripheral Sensory Neuropathy (Nervous system disorders) | 7 | 1
Syncope (Nervous system disorders) | 2 | 3
Anxiety (Psychiatric disorders) | 20 | 6
Depression (Psychiatric disorders) | 13 | 2
Insomnia (Psychiatric disorders) | 14 | 10
Dysuria (Renal and urinary disorders) | 6 | 3
Vaginal Haemorrhage (Reproductive system and breast disorders) | 6 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 12
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 13 | 6
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 12 | 2
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 5
Erythema (Skin and subcutaneous tissue disorders) | 5 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9 | 3
Night Sweats (Skin and subcutaneous tissue disorders) | 6 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 10 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 4
Rash (Skin and subcutaneous tissue disorders) | 37 | 11
Deep Vein Thrombosis (Vascular disorders) | 5 | 1
Hypertension (Vascular disorders) | 11 | 6
Hypotension (Vascular disorders) | 18 | 6
Abdominal pain lower (Gastrointestinal disorders) | 4 | 3
Enterococcal bacteraemia (Infections and infestations) | 3 | 4
Staphylococcal bacteraemia (Infections and infestations) | 6 | 1
Urinary tract infection enterococcal (Infections and infestations) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 9 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 6
Rash erythematous (Skin and subcutaneous tissue disorders) | 6 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No